CLINICAL TRIAL: NCT03043638
Title: Efficiency of Platelet-Rich Plasma (PRP) on Acellular Dermal Matrix Application With Coronally Advanced Flap in the Treatment of Multiple Adjacent Gingival Recessions:a Double-masked Randomized Controlled Clinical Trial
Brief Title: Efficiency of PRP on Acellular Dermal Matrix Application in the Treatment of Multiple Adjacent Gingival Recessions
Acronym: PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, PELİN GÖKALP, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03/2007-28
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-01

CONDITIONS: Gingival Recession, Generalized
Keywords: multiple adjacent gingival recessions; platelet rich plasma; acellular dermal matrix; coronally advanced flap; gingival recession; root coverage; clinical attachment level
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAF+ADM+PRP (Experimental): Surgery will include Coronally advanced flap(CAF) plus acellular dermal matrix (ADM) combined with platelet rich plasma (PRP)
  Interventions: Procedure: CAF+ADM+PRP
- CAF+ADM (Active Comparator): Surgery will include only Coronally advanced flap CAF technique including ADM placement without PRP
  Interventions: Procedure: CAF+ADM

INTERVENTIONS:
Procedure: CAF+ADM+PRP — CAF+ADM+PRP group treated with coronally advanced flap technique including ADM placement, In CAF+ADM+PRP group, ADM was hydrated in the platelet-poor plasma (PPP) and the PRP was applied to surgical sites prior to final suturing.
  Arms: CAF+ADM+PRP
Procedure: CAF+ADM — CAF+ADM group treated with coronally advanced flap technique including ADM placement without PRP application
  Arms: CAF+ADM

SUMMARY:
The aim of this study was to evaluate the effectiveness of platelet rich plasma (PRP) combined with coronally advanced flap plus acellular dermal matrix application (CAF+ADM) in the treatment of multiple adjacent gingival recessions (MAGRs).

12 patients with 84 Miller Class I or II recession defects were participated. Sites were randomly assigned into CAF+ADM+PRP or CAF+ADM groups. Gingival recession depth (GRD), recession width (GRW), width of keratinized tissue (WKT), creeping attachment (CRA), root coverage (RC) as well as plaque index, gingival index, probing depth (PD), and clinical attachment level (CAL) were recorded at baseline and 3rd,6th and 12th months postoperatively. The data were analyzed statistically.

DETAILED DESCRIPTION:
Several methods have been demonstrated for the treatment of gingival recession defects with the use of PRP. In an 8-month randomized controlled trial, it was reported that there was no significant difference between PRP and CTG treated groups in terms of root coverage of Miller Class 1 or II buccal recession defects. However, in the same study contour and texture of soft tissue showed valuable enhancement in PRP group. The use of PRP together with ADM in the treatment of MAGRs may alleviate the need for autogenous donor tissue. Shepherd et al. compared coronally positioned tunnel technique and ADM application with and without PRP for the treatment of single gingival recession defects and reported no statistically significant root coverage difference between groups.

Although there are numerous root coverage procedures to treat the conditions, predictable coverage of multiple adjacent gingival recessions still remains a challenge for the clinician. The aim of this randomized, controlled, clinical trial was to compare the CAF plus ADM application together with and without PRP to determine whether the PRP provided an advantage in terms of gaining coverage of deep and wide recession defects in the treatment of MAGRs.

In the present study, using a controlled blinded split-mouth design, 14 patients with multiple Miller Class I or II adjacent recession defects ≥ 3mm deep on bilateral operation sites were randomly operated either with CAF+ADM+PRP or only CAF+ADM as test and control groups respectively. Two patients who failed to return for all postoperative visits were exited from the study.

Finally12 patients who had adjacent Miller Class 1 or II (Miller) recession defects ≥ 3mm deep on non-molar teeth in the same dental arch at least two bilateral site, underwent through root coverage surgery and were followed for 12 months. The study sample consisted of 84 teeth associated with total of 12 patients; seven patients each showing a pair of three teeth, four patients each showing a pair of four teeth, and one patient showing a pair of five teeth with adjacent multiple recessions deep on the buccal aspect of each tooth. The treated teeth were 26 incisors, 24 canines and 34 first premolars. Standardized radiographs were taken to evaluate the interproximal alveolar bone level. At baseline, 3, 6 and 12 months after the surgeries; Miller classification of the recession defect (Miller, 1985), plaque index (PI) (Silness and Loe, 1964), gingival index (GI) (Loe, 1967) probing depth (PD), clinical attachment level(CAL), Probing depth(PD), gingival margin (GM), Gingival recession width (GRW) were recorded. The pre-surgical evaluation included an analysis of the patient's tooth brushing technique and habits. At the teeth showing gingival recessions, a coronally directed roll technique using a soft toothbrush was indicated to minimize the tooth brushing trauma to the gingival margin. Pre-surgical therapy included scaling, root planning, polishing and general oral hygiene instruction. All surgical procedures were performed with Coronally Advanced Flap technique.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of the presence of at least three multiple adjacent Miller class I or II recessions on both sides of the same maxillary or mandibular arch
2. must be able to have 2 mm-high keratinized tissue apical to the root exposures;
3. must be able to have no systemic diseases that could influence the outcome of the therapy;
4. must be able to have a full-mouth plaque score of 20% (O'Leary et al. 1972);
5. must be non-smoker;
6. must be not pregnant.

Exclusion Criteria:

* debilitating systemic or infectious diseases (human immunodeficiency virus or hepatitis) -- -any disease that significantly affects the periodontium;
* known allergy to any of the materials used in the study; requirement for antibiotic prophylaxis;
* taking medications known to interfere with periodontal health and healing not detectable cemento-enamel junction (CEJ);
* restorations or caries at the recession site;
* failure to maintain an oral hygiene level ≥80% plaque-free surfaces; pregnancy or lactation; use of tobacco products; alcohol abuse;
* a previous periodontal surgery at the recession site and failure to complete the informed consent.

Ages: 34 Years to 57 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-07-01 (Actual); Primary Completion 2011-06-20 (Actual); Study Completion 2011-06-20 (Actual)

PRIMARY OUTCOMES:
Root coverage (RC) | The change in RC at 3rd month to 12th month
  The percentage of root coverage (RC) was calculated as ([GRD preoperation - GRD postoperation] / GRD preoperation) x 100%.

SECONDARY OUTCOMES:
Gingival recession depth (GRD) | Baseline, 3,6 and 12 months after periodontal surgery
  The GRD was measured from the CEJ to the GM. PD, CAL and GRD were measured at the same reference points.
recession width (GRW) | Baseline, 3,6 and 12 months after periodontal surgery
  Gingival recession width (GRW) was measured with perpendicular positioning of the periodontal probe to the cemento-enamel junction, the distance between the top of the papilla at the mesial and distal aspect of the tooth was recorded.
width of keratinized tissue (WKT) | Baseline, 3,6 and 12 months after periodontal surgery
  Width of keratinized tissue (WKT) was measured at the mid-buccal point from the mucogingival junction (MGJ) to the free GM by a digital caliper.
plaque index(PI) | Baseline, 3,6 and 12 months after periodontal surgery
  plaque index were calculated as a sum of mean scores by each examined tooth divided by the number of evaluated teeth. A mean of all measurements for each patient was considered.
gingival index | Baseline, 3,6 and 12 months after periodontal surgery
  gingival index were calculated as a sum of mean scores by each examined tooth divided by the number of evaluated teeth. A mean of all measurements for each patient was considered.
probing depth | Baseline, 3,6 and 12 months after periodontal surgery
  PD was measured at three points (mesio-buccal, midbuccal, and disto-buccal) on the individual elastomeric stent and calculated as the distance between gingival margin (GM) and the bottom of the sulcus.

CONTACTS AND LOCATIONS:
Overall Officials: Pelin Gokalp, Principal Investigator — Gazi University

IPD SHARING:
Plan to Share IPD: Yes
When needed data can be shared via email.

REFERENCES:
- [Background] Shepherd N, Greenwell H, Hill M, Vidal R, Scheetz JP. Root coverage using acellular dermal matrix and comparing a coronally positioned tunnel with and without platelet-rich plasma: a pilot study in humans. J Periodontol. 2009 Mar;80(3):397-404. doi: 10.1902/jop.2009.080438. PMID 19254123
- [Derived] Cetiner D, Gokalp Kalabay P, Ozdemir B, Cankaya ZT. Efficiency of platelet-rich plasma on acellular dermal matrix application with coronally advanced flap in the treatment of multiple adjacent gingival recessions: A randomized controlled clinical trial. J Dent Sci. 2018 Sep;13(3):198-206. doi: 10.1016/j.jds.2017.11.002. Epub 2018 Feb 3. PMID 30895121